CLINICAL TRIAL: NCT05299840
Title: Impact of Using the Oncogramme® Device to Select the First Line of Treatment (Chemotherapies +/- Targeted Therapies) for Patients With Metastatic Colorectal Cancer on Progression-free Survival, Treatment Costs, Efficiency and Quality of Life Compared to Usual Patient Care.
Brief Title: Impact of Using the Oncogramme® Device to Select the First Line of Treatment for Patients With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oncomedics (Industry)
Collaborators: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ONCOG
Record Dates: First submitted 2022-03-10; First posted 2022-03-29 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oncogramme group (Experimental): The oncologist has access to the results of the Oncogramme® Device and decides on the treatment according to the recommendations of the Oncogramme® Device
  Interventions: Diagnostic Test: Oncogramme results available
- Control group (Other): The oncologist does not have access to the results of the Oncogramme® Device and decides on the treatment according to the standard of care.
  Interventions: Diagnostic Test: Oncogramme results unavailable

INTERVENTIONS:
Diagnostic Test: Oncogramme results available — in vitro analysis of each patient's tumor cells in order to compare the responses of the tumor cells to the different molecules and therapeutic combinations available
  Arms: Oncogramme group
Diagnostic Test: Oncogramme results unavailable — in vitro analysis of each patient's tumor cells in order to compare the responses of the tumor cells to the different molecules and therapeutic combinations available
  Arms: Control group

SUMMARY:
Colorectal cancer is the 2nd leading cause of cancer death in France. Its incidence is nearly 45,000 new cases per year in 2017, with an estimated 5-year survival of 63% in 2015. Metastases are seen in 40-60% of colorectal cancer cases. The 5-year survival rate ranges from 5% to 15% for patients with widespread metastatic disease.

Two types of treatments are used to treat colon cancer: surgery and medication protocol (chemotherapeutic drugs and targeted therapies). These treatments can be used alone or in combination.

The current choice of a first line of chemotherapy is left to the practitioner's discretion, after consultation with a multidisciplinary consultation meeting. The choice of treatment(s) depends on official recommendations and is based on the results of clinical trials conducted on large populations, and takes into account the toxicities of the therapies used and the general condition of the patients. The therapeutic combinations for colorectal cancers are therefore multiple. However, to date, no consensus has been reached to ensure that each patient is treated effectively and as a unique case.

Today, functional sensitivity tests offer the possibility for patients to be offered a personalized treatment against cancer. This is the case of the Oncogramme® device developed by Oncomedics, which is the first functional sensitivity test dedicated to oncology in Europe. It is based on an in vitro analysis of each patient's tumor cells in order to compare the responses of the tumor cells to the different molecules and therapeutic combinations available (chemotherapy ± targeted therapy). This response, translated into a tumor-specific sensitivity profile, can be used by the medical team to determine the most appropriate treatment for the patient. This test is therefore likely to improve the benefit-risk ratio of a chemotherapy treatment in colorectal cancer by allowing the medical team to select, among the treatments deemed effective, the one that will be the most effective on the tumor and possibly with the least side effects.

The hypothesis of this study is that the personalization of treatments (by chemotherapy associated or not with targeted therapies) proposed by the Oncogramme®-colorectal device would allow to promote the best possible clinical response, to limit the side effects and ultimately to improve the survival and the quality of life of the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Patient with suspected mCRC (synchronous or metachronous metastases (only if biopsy is required as part of routine care))
* Patient eligible for standard systemic chemotherapy (multidrug therapy such as FOLFOX, FOLFIRI, FOLFIRINOX, combined or not with anti- EGFR or anti-VEGF targeted therapies adapted to BRAF and RAS expression)
* colorectal adenocarcinoma histologically proven
* At least one measurable metastasis according to RECIST v1.1
* Chemotherapy for curative or palliative purposes
* Oncograms® can be performed
* WHO score ≤ 2
* Life expectancy > 3 months
* neutrophils > 1500/mm3, platelets > 100 000/mm3, Hb > 9 g/dL
* Total bilirubin < 25 μmol/L, aspartate aminotransferase < 5 ULN (upper limits of normal), alanine aminotransferase < 5 ULN, alkaline phosphatase < 5 ULN, prothrombin rate > 60%, proteinuria < 1 g/24h
* No prior chemotherapy except peri-operative or adjuvant chemotherapy stopped more than 6 months ago
* Creatinine clearance > 50 mL/min according to MDRD formula
* Patient affiliated to a social security scheme
* Information to the patient and signature of the informed consent form.

Exclusion Criteria:

* Patients eligible for curative treatment (surgical and/or percutaneous) after discussion in multidisciplinary consultation meeting (isolated class I liver metastases)
* Patients with metachronous metastases not requiring biopsy as part of their standard management.
* Myocardial infarction, severe/unstable angina, coronary artery bypass grafting, New York Heart Association (NYHA) class II, III, or IV congestive heart failure, stroke, or transient ischemic attack within 6 months prior to inclusion
* HTA not controlled by medical treatment (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg)
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active gastrointestinal bleeding in the 6 months preceding the start of treatment
* Active peptic ulcer
* Deep wound or bone fracture not resolved within 3 months
* Major abdominal or extra-abdominal surgical procedure (except diagnostic biopsy or implantable site placement)
* Irradiation within 4 weeks prior to the start of treatment
* Transplant patients, HIV-positive, or other immunodeficiency syndromes
* Previous chemotherapy (except peri-operative or adjuvant chemotherapy discontinued more than 6 months ago)
* Any progressive disease not balanced during the last 6 months: hepatic insufficiency, renal insufficiency, respiratory insufficiency
* Peripheral neuropathy > 1 (CTCAE Common terminology criteria for adverse eventsv5.0)
* Patient with interstitial lung disease or pulmonary fibrosis
* History of chronic diarrhea or inflammatory disease of the colon or rectum, or occlusion or sub-occlusion unresolved with symptomatic treatment
* History of malignancy within the last 5 years except for properly treated non-metastatic colon cancer, basal cell skin carcinoma or carcinoma in situ of the uterine cervix
* Patient already included in another therapeutic trial with an investigational treatment or who has been out of a trial for less than 6 months
* Any specific contraindication or known allergy to the drugs used in the study.
* Known dihydropyrimidine dehydrogenase deficiency
* QT/QTc interval > 450 ms for men and > 470 ms for women
* Kalemia (K+) < LIN (lower limit to normal), magnesemia (Mg2+)< LIN, calcemia (Ca2+)< LIN
* Lack of effective contraception (at least 2 different means) in patients (male or/and female) of childbearing age, or for females, 12 months of confirmed amenorrhea, pregnant or lactating woman, woman of childbearing age who has not performed a pregnancy test (serum test)
* Persons deprived of liberty or under guardianship
* Impossible to undergo the medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 12 months
progression-free survival | 24 months

SECONDARY OUTCOMES:
Objective response rates | 12 months
  Sum of complete and partial remission rates measured according to RECIST v1.1
Objective response rates | 24 months
  Sum of complete and partial remission rates measured according to RECIST v1.1
Response time | 12 months
  Time from first recognition of response to first recognition of progress
Rate of treatment change due to tumor progression | 2 months
Overall survival | 24 months
Diagnostic performance of the Oncogramme device | 12 months
  Calculation of the sensitivity, specificity, and predictive Values of the Oncogramme device
Budget impact | 12 months
  Calculation of incremental and avoided costs per patient
Quality of life of patients | 12 months
  measured using EORTC core quality of life questionnaire (QLQ-C30)
Quality of life of patients | 24 months
  measured using EORTC core quality of life questionnaire (QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Perrier, M.D, Principal Investigator — Hopital Saint Joseph Marseille
Locations (1):
- Hôpital Saint Joseph Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No